CLINICAL TRIAL: NCT06521437
Title: Hippocampal Network Function in Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB23-1089
Record Dates: First submitted 2024-07-08; First posted 2024-07-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Mesial Temporal Lobe Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experiment 1 (Experimental): Subjects will be tested for baseline performance on a memory task while in an MRI scanner and with scalp EEG. Subjects will then receive multiple sessions, of repetitive transcranial magnetic stimulation. Post-treatment, baseline assessments will be repeated. Overall study period per subject: 2 months
  Interventions: Device: TMS targeting the hippocampus indirectly via its network

INTERVENTIONS:
Device: TMS targeting the hippocampus indirectly via its network — Subjects will receive high-frequency repetitive TMS to a parieto-occipital location defined in each subject based on high resting-state fMRI connectivity with the hippocampus at baseline

SUMMARY:
The aim of this pilot study is to understand hippocampal network function in mesial temporal lobe epilepsy (MTLE) and to test whether transcranial magnetic stimulation (TMS) targeting the network of the hippocampus can change hippocampal-dependent memory task performance and epileptic activity in people with (MTLE). Positive findings would implicate the hippocampal network as a source of these typical primary MTLE symptoms.

Subjects with a primary diagnosis of MTLE will be enrolled in a non-randomized, non-blinded pilot experiment to test target engagement and preliminary efficacy of a novel neurostimulation approach targeting the hippocampal network. At baseline, subjects will undergo neurocognitive testing for hippocampal-dependent memory and functional magnetic resonance imagining (fMRI) neuroimaging assessment of brain structure and task-dependent activity. They will also receive scalp-electroencephalography (EEG) to measure interictal epileptiform discharge (IED) frequency at baseline, and will complete a seizure diary for one month. They will then receive high-frequency repetitive TMS targeting an area of parieto-occipital cortex defined based on fMRI connectivity with the hippocampus measured at baseline. The baseline assessments will then be repeated, using an alternate form of the memory test. The investigators will analyze changes from baseline in memory task performance, fMRI activity of the hippocampal network, IED frequency, and reported seizure frequency.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate hippocampal network dysfunction associated with mesial temporal lobe epilepsy (MTLE) and to examine whether network-targeted transcranial magnetic stimulation (TMS) can affect hippocampal connectivity, cognitive performance, and epileptic activity observed in adult subjects with MTLE.

Subjects will be recruited through the University of Chicago Medicine Comprehensive Epilepsy Center and other local epilepsy centers. Subjects will complete up to 8 experimental sessions (1 baseline experiment/assessment, up to 5 TMS sessions, up to 2 post-treatment experiments/assessments), spread over a two-month period. During the baseline and post-treatment sessions, subjects will undergo electroencephalography (EEG) and functional magnetic resonance imaging (fMRI). EEG will be utilized to examine interictal epileptiform discharge (IED) frequency at rest as well as task-related neural activity recorded from non-invasive scalp EEG electrodes at locations conforming to the International 10-20 positioning system with additional anterior temporal electrodes. MRI scanning procedures will take approximately 45 minutes and include native anatomical (MP-RAGE) as well as functional (EPI) sequences to assess hippocampal network function and task-related activity. During both, the EEG and MRI procedures, subjects will perform a memory task.

One month following the baseline session, subjects will return to the lab for up to 5 TMS intervention sessions. During the one-month period preceding TMS, subjects will complete a daily seizure diary to track baseline seizure frequency prior to the intervention. TMS parameters are determined based on the allowable dosage of TMS delivery, calculated based on published standards for experimental TMS protocols, and in accordance with standard operating procedures for TMS. Subjects will receive brief (~2 to 40s) trains of repetitive TMS with long (>10s) inter-train intervals. Each train of repetitive TMS will include between 20 and 40 individual pulses delivered at frequencies hypothesized to have different effects on memory (e.g., in the theta range). Individual pulse intensity will be calibrated using the motor-threshold method. Post-treatment sessions will once again comprise EEG and fMRI procedures as described above. Following the post-treatment sessions, subjects will continue to complete a daily seizure diary for the next 30 days to track any changes to seizures following treatment. Pre- and post-stimulation data will be compared to assess effects of the intervention on memory performance, hippocampal network function, and epileptic activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of (pharmacoresistant) MTLE
* Age 18+ years old
* Native English speakers
* Normal or corrected-to-normal near and far vision
* Stable antiepileptic drugs (AED) regimen (unchanged for at least 1 month)

Exclusion criteria:

* Diagnosis of neurological illness other than MTLE
* Taking drugs that impair cognition other than anticonvulsive medication for the treatment of MTLE (e.g., antipsychotics or psychostimulants).
* Children under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Epileptic activity (IEDs) | Measured at baseline and 1 day after stimulation
  Scalp EEG is used to measure IEDs, identified via clinical assessment and quantified

SECONDARY OUTCOMES:
Memory task performance | The memory task is administered at baseline and 1 day after the last stimulation session. Recall will be measured approximately 15 minutes after seeing the word pairs.
  Subjects memorize word pairs and then attempt to recall the missing word given one item from each pair after a delay. Total number of words pairs recalled will be measured.
fMRI connectivity of the hippocampal network | First day of study (baseline session) and 1 day after last stimulation session.
  Subjects will undergo MRI neuroimaging assessment of brain structure and resting-state function. The correlation between the hippocampus and parietal cortex will be measured.
Seizure frequency reported in seizure diary | From the baseline session to 30 days following the post-treatment sessions
  Subjects will complete an online seizure diary daily. Number of daily seizures reported will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Voss, PhD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552